CLINICAL TRIAL: NCT06139575
Title: Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Radiation Dosimetry and Preliminary Efficacy of Lutetium Lu 177 JH020002 Injection in Patients With Advanced Prostate Cancer
Brief Title: Phase 1/2 Clinical Study of Lutetium Lu 177 JH020002 Injection in Patients With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bivision Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JH020002-01C
Record Dates: First submitted 2023-11-09; First posted 2023-11-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lutetium Lu 177 JH020002 Injection (Experimental)
  Interventions: Drug: Lutetium Lu 177 JH020002 Injection

INTERVENTIONS:
Drug: Lutetium Lu 177 JH020002 Injection — Patients will receive Lutetium Lu 177 JH020002 Injection every 6 weeks for a maximum of 6 doses. Doses range between 1.85 and 8.88 GBq (50-240 mCi)

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics, radiation dosimetry, and preliminary efficacy of Lutetium Lu 177 JH020002 Injection in adult patients with advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are required to get informed consent prior to the trial and sign a written informed consent form voluntarily.
* Male, age ≥18 years.
* ECOG score 0 - 2.
* Must have a life expectancy >6 months.
* Histologically and/or cytologically confirmed adenocarcinoma of the prostate (except for those with neuroendocrine or small cell prostate cancer clinical features).
* Participants must have a castrate level of serum/plasma testosterone (< 50 ng/dl, or < 1.7nmol/L).

Exclusion Criteria:

* Diagnosed with other malignancies, apart from: adequately treated skin basal cell carcinoma or superficial bladder cancers from which the patient has been disease-free for more than 3 years as confirmed by a physician.
* Participants with a history of central nervous system (CNS) metastases who are neurologically unstable, symptomatic, or receiving corticosteroids for the purpose of maintaining neurologic integrity.
* Previous treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation <6 months prior to date of first administration of investigational drug.
* Previous PSMA-targeted radioligand therapy.
* Previous radiotherapy for prostate cancer within 4 weeks prior to date of first administration of investigational drug.
* Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy, poly adenosine diphosphate-ribosyl polymerase inhibitors (PARPi) or biological therapy within 4 weeks prior to date of first administration of investigational drug.
* Must not take part in other investigational therapies within 4 weeks prior to date of first administration of investigational drug.
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) (Phase 1) | Up to 2 years follow up
  Incidence of adverse events, serious adverse events, and clinical laboratory abnormalities defined as dose-limiting toxicities (DLTs).
Maximum Tolerated Dose (MTD) (Phase 1) | Up to 2 years follow up
  The maximum tolerated dose is among the explored dose levels.
Recommended Phase 2 Dose (RP2D) (Phase 1) | Up to 2 years follow up
  To identify the expansion phase dose of Lutetium Lu 177 JH020002 Injection.
PSA response rate | Up to 3 years follow up
  PSA response rate is the proportion of PSA responders, defined as a participant who has achieved PSA decrease of >= 50% from baseline that is confirmed by a second consecutive PSA measurement >= 4 weeks later. Determination of response status will be based on PCWG3 recommendations.

SECONDARY OUTCOMES:
Radiation Dosimetry | Up to 2 years follow up
  Absorbed dose estimated in organs and tumor lesions.
Maximum plasma concentration (Cmax) | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Time to maximum plasma concentration (Tmax) | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Terminal elimination half-life (t1/2) | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Total systemic clearance (CL) | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC0-t) | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC0-inf) | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Volume of distribution (Vz) during the terminal phase following intravenous elimination | Up to 2 years follow up
  Pharmacokinetics (PK) characterization of Lutetium Lu 177 JH020002.
Radiographic Progression-free Survival (rPFS) | Up to 3 years follow up
  Radiographic progression free survival (rPFS) is defined as the time of radiographic progression by Prostate Cancer Working Group 3 (PCWG3)-modified RECIST V1.1.
Disease control Rate (DCR) | Up to 3 years follow up
  Disease control rate (DCR) is defined as the proportion of participants with best overall response of complete response or partial response or Stable disease in soft tissue according to PCWG3 modified RECIST 1.1.
Duration of Response (DoR) | Up to 3 years follow up
  Duration of response (DOR) is defined as the duration of time between the date of first documented response (CR or PR) in soft tissue as per BIRC and according to PCWG3 modified RECIST 1.1, and the date of first documented progression or death due to any cause.
Time to First Subsequent Therapy (TFST) | Up to 3 years follow up
  Time to First Subsequent Therapy (TFST) is defined as the time from the date of first administration of investigational drug to the date of the first subsequent therapy of the prostate cancer.
Overall Survival (OS) | Up to 3 years follow up
  Overall survival (OS) is defined as the time from the date of first administration of investigational drug to the date of death due to any cause.
Time to Symptomatic Skeletal Event (TTSSE) | Up to 3 years follow up
  Time to a first symptomatic skeletal event (TTSSE) is defined as date of first administration of investigational drug to the date of first new symptomatic pathological bone fracture, spinal cord compression, tumor-related orthopedic surgical intervention, requirement for radiation therapy to relieve bone pain or death from any cause, whichever occurs first.
Incidence and severity of Adverse Events (AEs) and Serious Adverse Event (SAEs) | Up to 3 years follow up
  Analysis of frequencies and severity for Adverse Events (AEs) and Serious Adverse Event (SAEs), through the monitoring of relevant clinical and laboratory safety parameters.
Objective Response Rate (ORR) (Phase 2) | Up to 2 years follow up
  Proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on the Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria response for patients with measurable disease at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Bivision Pharmaceuticals, Inc., Study Director — Bivision Pharmaceuticals, Inc.
Locations (13):
- China (13):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Huazhong University of Science and Technology Tongji Medical College Affiliated Union Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Wuxi, Jiangsu
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Bivision Pharmaceuticals, Inc. is committed to sharing with qualified external researchers access to patient-level data. These sharing requests are reviewed and approved by Bivision Pharmaceuticals, Inc subject to certain criteria and conditions. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.